CLINICAL TRIAL: NCT03296644
Title: "Evaluation of Treatment Effects of Two Different Fixed Functional Appliances in Patients With Class II Div 1 Malocclusion Using CBCT- A Randomized Controlled Clinical Study"
Brief Title: Comparison of Treatment Effects of PowerScope2 and Forsus Using CBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sonal ortho
Record Dates: First submitted 2017-09-09; First posted 2017-09-28 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PowerScope2 group (G1) (Active Comparator): Class II correction using PowerScope2
  Interventions: Device: Class II correction using PowerScope2
- Forsus group (G2) (Active Comparator): Class II correction using Forsus
  Interventions: Device: Class II correction using Forsus

INTERVENTIONS:
Device: Class II correction using PowerScope2
  Arms: PowerScope2 group (G1)
Device: Class II correction using Forsus
  Arms: Forsus group (G2)

SUMMARY:
The main objective of this prospective, controlled clinical study is:

1. To compare the treatment effects of PowerScope2 and Forsus Fatigue Resistant Device in patients with Class II divison1 malocclusion.
2. To compare the treatment effects of PowerScope2 and Forsus Fatigue Resistant Device with the control group.

The null hypothesis for this study is that Forsus and PowerScope2 are equally effective in the treatment of ClassII div1 malocclusion.

DETAILED DESCRIPTION:
Class II malocclusion is one of the most frequent problems in orthodontics ,as it affects one third of patients seeking orthodontic treatment. McNamara reported mandibular retrusion as the most common characteristic of Class II malocclusion rather than maxillary prognathism. Functional orthopaedic appliances are widely used to treat Class II malocclusion in growing patients .Contrary to removable appliances, fixed devices do not require patient collaboration and can be worn in association with multibracket therepy, so that class II malocclusion can be corrected in a single phase treatment.

.Most popular flexible devices are the Jasper Jumper, Eureka spring, and the Forsus device (FRD)Forsus Fatigue Resistant Device [FRD]is a three piece (L pin module) or two-piece (EZ2 module) system, composed of a telescoping spring that attaches at upper first molar and a push rod linked to lower archwire, distal to either the canine or first premolar bracket. The FRD spring and rod create an equal and opposite force to maxillary and mandibular dentition.1The clinical application of the FRD was described by Vogt in 2006.PowerScope is one of the latest innovation in Class II correction developed by Dr. Andy Hayes. Inventors claims the following advantages of powerscope over other functional appliances. It is delivered as a one-size-fits-all appliance pre-assembled with attachment nuts for quick and easy chairside application .

The appliance is a wire-to-wire installation with attachments placed mesial to the first molar in the maxillary arch and distal to the canine of the mandibular arch. Internal NiTi spring mechanism delivers 260 gms of force for continous activation during treatment.

The dental, skeletal and soft tissue short-term effects of comprehensive fixed appliance treatment combined with ForsusTM in ClassII patients have been evaluated previously. However no previous study compared the posttreatment effects of PowerScope2TM and ForsusTM.The purpose of this controlled clinical study is to evaluate the treatment and posttreatment effects induced by PowerScope2 in growing patients with ClassII malocclusion and to compare it with Forsus(FRD) on CBCT.

The majority of the studies examined the changes of the upper airway through lateral cephalometric radiography. This method limited the accuracy of airway measurement since the two-dimensional (2D) images only allowed an anteroposterior dimension measurement in sagittal plane, and failed to provide a full-scaled view of the upper airway. Therefore, 3D evaluation of the upper airway in growing patients during fixed functional appliance treatment needs to be established .Cone beam computed tomography (CBCT) is an acceptable technique for 3D volumetric depiction and morphological evaluation of the upper airway using a lower-radiation method with a greater spatial resolution . It allows 3D registration of pre- and post-treatment data through identification of specific structures in the cranial base. Therefore, the changes of the upper airway before and after mandibular advancement can be precisely evaluated. As the patients involved in our research were underage, their normal development may affect on the upper airway morphology during the treatment period. Thus, an untreated control group is needed. In the present study, the control group was selected from records of patients with the same diagnosis who just began orthodontic treatment, and matches well with the post-treatment patients of fixed functional appliance group through age, sex and development condition strategy, so that effects of fixed functional appliance on the upper airway morphology can be evaluated.

MATERIALS AND METHODS- Ours is a prospective, non-pharmacological, double blind, randomized controlled clinical study to compare the treatment effects of two different fixed functional appliances, Forsus and PowerScope2. The present study will be conducted in the Department of Orthodontics and Dentofacial Orthopedics, PGIDS, Pt. B.D. Sharma University of Health Sciences, Rohtak.

Ethical clearance- The study will be carried out after the institutional approval for use in humans.

Source of data:- The sample size consists of 63 subjects who were selected from the patients attending regular OPD at the Department of Orthodontics and Dentofacial Orthopedics for orthodontic treatment.

TARGET SAMPLE SIZE Nearly 21 subjects per group and 63 in total should be an ideal sample size including 10% dropout for the proposed study to have a power of 90% and a standard error of significance to be 0.05.

INFORMED CONSENT OF THE PATIENT AND AGREEMENT TO BE RANDOMISED A valid, informed written consent of the patient or parent/ guardian and an agreement to be randomized was obtained from the patient before registering the patient in this clinical study. Patient or parent/ guardian was informed about all the theoretical risks and benefits of the intervention under test. Risks and hazards of radiation during CBCT were also explained to the patient.

INTERVENTION AND DESIGN OF STUDY

The main intervention in this clinical study is placement of 2 different fixed functional appliances after initial levelling and alignment of dental arches. The study consists of 3 groups with equal allocation of subjects in each group-

G1- This group received Powerscope2 appliance bilaterally G2-This group received Forsus bilaterally (as per size suitable for the individual.

G3-The control group wiil be selected from patients with same diagnosis who just began orthodontic treatment, and matches well with the post treatment patients of Powerscope2 and Forsus through age, sex and development condition.

Selection of subjects in intervention groups (patients meeting selection criteria)

Treatment with 0.022 MBT preadjusted edgewise appliance

Maxillary and mandibular arches will be stabilized with the help of 0.019" × 0.025" stainless steel wire, reverse torque will be introduced in the lower anterior segment and wires will be cinched back distal to 2ndmolars.

Patient were randomly allocated into 2 groups.

1 PowerScope2 (G1) 2. Forsus (G2)

Pretreatment diagnostic records including lateral cephalogram were taken. CBCT was taken before insertion and after removal of the fixed functional appliance.

Insertion of fixed functional appliance as per the group allocated. Regular follow up till the completion of functional phase of treatment will be done. Patients will undergo functional appliance phase till Class I molar relationship is achieved.

RANDOMISATION & ALLOCATION CONCEALMENT The subjects were randomly allocated by a sealed opaque envelope method. The study subjects were blinded regarding intervention group. Allocated appliance was inserted on the patient.

DATA COLLECTION AND CBCT ANALYSIS

The investigator recorded the patients' name, address and contact number. CBCT will be recorded before placement of fixed functional appliance and immediately after its removal in order to evaluate changes caused by the functional appliances.

To check patient comfort, all patients were given a questionnaire to investigate the patient's experiences with PowerScope2 and Forsus. The questionnaire was designed in English and then verbally translated into the patients and parents native language at the installation appointment though all the patients and their parents could read and understand it in English.

Prefunctional and postfunctional profile photographs of the treatment groups (G1 and G2) patients and those of control will be presented to 5 orthodontists, 5 patients, 5 parents and 5 laypersons.The raters will assess changes in facial appearance on a visual analog scale.

CBCT Data Acquisition The pre-treatment and post-treatment CBCT scans of two intervention groups (G1 & G2) and the CBCT of control group (G3) will be collected and analysed.

During CBCT scan, patients will be instructed to maintain an upright posture and natural head position. The CBCT scans will be performed at rest position of the tongue (tongue in contact with anterior palate without touching the anterior teeth) and maximum intercuspation. All of the scans will be performed by the same researcher.

DATA COLLECTION & INTERPRETATION Data will be collected, properly arranged and a CONSORT flow chart will be made to derive final sample size and calculate number of exclusions.

Statistical analysis:-The data recorded will be processed by standard statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients in active growth period
* Skeletal Class II malocclusion
* Normal or mildly prognathic maxilla
* Retrognathic mandible.
* Increased overjet, not less than 5 mm.
* Horizontal to average growth pattern
* Positive pretreatment visual treatment objective (VTO).
* Minimum crowding in dental arches.
* Treatment completed without any permanent teeth extracted (excluding third molars).

Exclusion Criteria:• Subjects with a history of orthodontic treatment

* Anterior open bite
* Severe proclination and crowding of anterior teeth
* Any systemic disease affecting bone and generalgrowth
* Vertical growth pattern
* Patient who fails to follow up or undergo complete treatment

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
mandibular length | 20 months
  changes in mandibular length after intervention
oropharyngeal volume | 20 months
  changes in oropharyngeal volumes after intervention
condylar changes | 20 months
  condylar changes after intervention
patient experiences | 20 months
  patient experiences with Forsus and PowerScope
pancherz analysis | 20 months
  pancherz analysis after intervention
soft tissue changes | 20 months
  soft tissue changes after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sonal Chowdhary, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol